CLINICAL TRIAL: NCT04807595
Title: A Multicenter Study to Estimate the Prevalence of HER2 Low and Describe the SoC, Treatment Patterns, and Outcome in Real-world Practice Among Unresectable and/or Metastatic Breast Cancer Patients With HER2-low Status - the RetroBC-HER2L Study
Brief Title: Estimation of the Prevalence of HER2 Low and Describe the SoC, Treatment Patterns, and Outcome in Real-world Practice Among Unresectable and/or Metastatic Breast Cancer Patients With HER2 Low Status
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: D9673R00004
Record Dates: First submitted 2021-03-18; First posted 2021-03-19 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: Metastatic breast cancer; Retrospective study; Epidemiology study; Human epidermal growth factor receptor 2 negative; Human epidermal growth factor receptor 2 low
MeSH Terms: conditions — Breast Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective cohort: Patients with confirmed diagnosis of HER2-neg, unresectable and/or mBC regardless of hormone status dating back from 31 December 2017 - but no older than 01 January 2015 - who progressed on any systematic anti-cancer therapy will be involved in this study.
  Interventions: Other: None (Observational study)

INTERVENTIONS:
Other: None (Observational study) — The data source for this project will be HER2 IHC historical scores, local lab rescoring of historical HER2 fixed tissue slides, independent central retesting or local lab retesting (under special occasions) of HER2 IHC status for enrolled patients who have available tissue, other biomarker testing results based on historical testing and/or testing of archived tissue samples when available, and curated patient-level data. Real-world data sources include electronic health records/electronic medical records (EHR/EMR) and biobank registries. Data from EHR/EMR sources will be curated. Biobank tissue for enrolled patients who have multiple samples available will be selected consecutively when possible and will start with the latest available samples then move backward in time.
  Other Names: Observational study

SUMMARY:
This is a worldwide, multicenter, non-interventional, retrospective study of patient medical records from metastatic breast cancer (mBC) patients previously identified as human epidermal growth factor receptor 2 negative (HER2-neg), regardless of hormone status.

DETAILED DESCRIPTION:
This is a worldwide, multicenter, non-interventional, retrospective study. The study will consist of 2 components. The first component involves local lab rescoring of qualified historical HER2 fixed tissue immunohistochemistry (IHC) stained slides (preferably using Ventana 4B5 assay) at sites (post-training) for mBC patients previously identified as HER2-neg, and independent central retesting of HER2 status using Ventana 4B5 assay for any enrolled patients with available archived tissue samples at designated central laboratories. Local lab rescoring and independent central retesting/local lab retesting will be conducted blinded of historical HER2 IHC scores.

The second component involves linking the rescored IHC status to the patient medical record either through registry databases or patient chart review. Such information will be used to describe the patient demographics, histopathological features, clinical presentation, and treatment patterns following mBC diagnosis, and clinical outcomes in real-world settings for all patients with HER2 scores of 0, >0 and < 1+, and 1+2+/ISH- (HER2 low). The clinicopathological and other relevant BC biomarker information will also be examined based on historical biomarker testing results and/or new testing conducted as part of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women:

   1. ≥ 18 years of age when consent provided for future sample and clinical data use - applicable for all countries participating in the study except Japan
   2. ≥ 20 years of age when consent provided for future sample and clinical data use - applicable for Japan only
2. Must have a histological or cytological confirmed diagnosis of unresectable or/and mBC between 01 January 2015 and 31 December 2017
3. Must have provided written consent allowing for data and samples to be used in the future and this study would be covered by the consent for future use. If the patient is deceased, a waiver may be accepted
4. Diagnosed as HER2-neg (HER2 IHC 0, 1+, 2+/ISH-), regardless of hormone status
5. Progressed on any systemic anti-cancer therapy (eg, endocrine therapy, chemotherapy, CDK4/6i, targeted therapies other than anti-HER2, or immunotherapy) in the metastatic setting
6. Must have historical HER2 fixed tissue IHC stained slides (preferably stained using Ventana 4B5 assay) in acceptable quality for accurate rescoring.

Exclusion Criteria:

1. Have a history of other malignancies, other than basal cell carcinoma of the skin and squamous cell carcinoma of the skin
2. Patients with historical HER2 status of IHC 2+/ISH+ or 3+, or HER2 amplified.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be eligible for study inclusion if their mBC diagnosis date is between 01 January 2015 and 31 December 2017 (dating back from 31 December 2017 but no older than 01 January 2015).
Sampling Method: Non-Probability Sample
Enrollment: 798 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Prevalence/Incidence of HER2 low among HER2-neg mBC patients, based on rescoring of historical HER2 fixed tissue IHC stained slides by Ventana 4B5 assay | Retrospective: From 01 January 2015 to 31 December 2020
  To describe the overall prevalence and disease burden of HER2 low (IHC 1+, 2+/ISH-) among unresectable and/or mBC patients identified as HER2-neg, based on rescoring of historical HER2 fixed tissue IHC stained slides by Ventana 4B5 assay. The prevalence of HER2 low (IHC 1+, 2+/ISH-) at unresectable/metastatic BC diagnosis, determined based on rescoring of historical HER2 IHC slides locally, among patients confirmed to be HER2-neg (HER2 IHC zero and HER2 IHC 1+ and 2+/ISH-) by rescoring of historical HER2 IHC slides, will be calculated by the following, based on the re-established HER2 status determined for each patient:
  Prevalence of HER2 low = (Number of patients with HER2 low)/(Total number of HER2 negative patients )
Disease outcome: Time to first subsequent treatment (TFST) | Retrospective: From 01 January 2015 to 31 December 2020
  To compare TFST between HER2 low BC patients and the HER2 IHC zero patient population. TFST is defined as the length of time from the initiation of treatment to the initiation of the patient's next systemic treatment.
Disease outcome: Time to treatment failure (TTF) | Retrospective: From 01 January 2015 to 31 December 2020
  To compare TTF between HER2 low BC patients and the HER2 IHC zero patient population. TTF is defined as the length of time from initiation of treatment to premature discontinuation.
Disease outcome: Overall survival (OS) | Retrospective: From 01 January 2015 to 31 December 2020
  To compare OS between HER2 low BC patients and the HER2 IHC zero patient population. OS is defined as the length of time from the initiation of treatment that patients are still alive.

SECONDARY OUTCOMES:
Clinicopathological characteristics in patients with HER2 low BC | Retrospective: From 01 January 2015 to 31 December 2020
  HER2 low disease will be assessed using descriptive statistics of histopathological and clinicopathological characteristics. A comparison will be made with the HER2 IHC zero patient population.
Concordance of HER2 rescore with historical HER2 score | Retrospective: From 01 January 2015 to 31 December 2020
  The concordance between historical HER2 IHC scores and local lab rescoring in the HER2-neg region (IHC score zero, 1+, and 2+) will be characterized.
  The concordance between historical scoringHER2 IHC scores and independent central retesting of HER2 IHC status in the HER2-neg region will be assessed using Cohen's Kappa statistics to assess agreement beyond chance alone. By convention, Kappa equal or greater than 0.8 is often considered almost perfect agreement, Kappa between 0.8 and 0.6 is considered substantial agreement.
Prevalence of HER2 low among unresectable and/or mBC patients identified as HER2-neg based on other IHC assays | Retrospective: From 01 January 2015 to 31 December 2020
  To describe HER2 low prevalence among unresectable and/or mBC patients identified as HER2-neg based on other IHC assays, compared with Ventana 4B5 assay.
Prevalence of HER2 low in HR-positive and HR-negative population | Retrospective: From 01 January 2015 to 31 December 2020
  The overall prevalence of HER2 low among unresectable and/or mBC patients identified as HER2-neg, regardless of assays used, will be summarized descriptively for HR-positive and HR-negative population, respectively.

CONTACTS AND LOCATIONS:
Locations (13):
- Research Site, Pittsburgh, Pennsylvania, United States
- Research Site, Melbourne, Australia
- Research Site, Montreal, Quebec, Canada
- Research Site, Clermont-Ferrand, France
- Research Site, Erlangen, Germany
- Research Site, Milan, Italy
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Isehara
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- Research Site, Seoul, South Korea
- Research Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Viale G, Basik M, Niikura N, Tokunaga E, Brucker S, Penault-Llorca F, Hayashi N, Sohn J, Teixeira de Sousa R, Brufsky AM, O'Brien CS, Schmitt F, Higgins G, Varghese D, James GD, Moh A, Livingston A, de Giorgio-Miller V. Retrospective study to estimate the prevalence and describe the clinicopathological characteristics, treatments received, and outcomes of HER2-low breast cancer. ESMO Open. 2023 Aug;8(4):101615. doi: 10.1016/j.esmoop.2023.101615. Epub 2023 Aug 8. PMID 37562195
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9673R00004&attachmentIdentifier=a54cdd1a-fd11-485d-bf1a-d07970630464&fileName=D9673R00004_CSR_Synopsis_Redacted.pdf&versionIdentifier=